CLINICAL TRIAL: NCT00135408
Title: Randomized, Double-Blind, Placebo-Controlled Phase II Study Comparing the Safety of MDX-010 (BMS-734016) Administered With or Without Prophylactic Oral Budesonide (Entocort EC) in Patients With Previously Treated Unresectable Stage III or IV Malignant Melanoma
Brief Title: A Study of MDX-010 (BMS-734016) Administered With or Without Prophylactic Oral Budesonide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Medarex (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CA184-007
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Malignant Melanoma
Keywords: Unresectable Stage III or IV Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Ipilimumab+ Placebo
- A2 (Active Comparator)
  Interventions: Drug: Ipilimumab+ Budesonide

INTERVENTIONS:
Drug: Ipilimumab+ Placebo — Solution, Intravenous, 10 mg/kg, 3 weeks, 12 - 48 weeks depending on the response.
  Other Names: BMS-734016; (MDX-010)
  Arms: A1
Drug: Ipilimumab+ Budesonide — Solution/Capsule, Intravenous/Oral, 10 mg/kg + 9 mg, 3 weeks (Ipilimumab) + once daily until week 16 (Budesonide), 12 - 48 weeks depending on the response.
  Other Names: BMS-734016; (MDX-010)
  Arms: A2

SUMMARY:
The purpose of the study is to determine Efficacy, Safety and Tolerability of MDX-010 (BMS-734016) administered with or without Prophylactic Oral Budesonide.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of unresectable Stage III or IV malignant melanoma (excluding ocular melanoma)
* Flexible Sigmoidoscopy and colonic biopsy required

Exclusion Criteria:

* Patients with active, untreated central nervous system metastasis. Patients with autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2005-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Rate of Grade 2,3,4 Diarrhea - patients on study drug.

SECONDARY OUTCOMES:
Safety monitored w/follow-up period. Assess Best Objective response, Disease control rate, progression free survival, overall survival, duration/best objective response, Time/best objective response. PK, immunogenicity & pharmacodynamic analysis | at Week 24

CONTACTS AND LOCATIONS:
Locations (10):
- United States (4):
  - Los Angeles, California
  - San Francisco, California
  - Charlotte, North Carolina
  - Seattle, Washington
- Canada (2):
  - Local Institution, Kitchener
  - Local Institution, Moncton
- Local Institution, Tel Aviv, Israel
- Local Institution, Forlì, Italy
- Local Institution, Lima, Peru
- Local Institution, Hull, United Kingdom

REFERENCES:
- [Derived] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx